CLINICAL TRIAL: NCT05113212
Title: Randomized, Prospective, Descriptive and Comparative Clinical Study of Macular Grasping Damage in Patients Undergoing Pars Plana Vitrectomy and Peeling of the Internal Limiting Membrane, Operated by Traditional Microscope or NGENUITY® 3D Visualization System With Heads-up Display System. A Pilot Study.
Brief Title: Damages From Macular Grasping During Vitrectomy Comparing Traditional and 3D Microscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Rita Daniele, MD (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor-Investigator, Anna Rita Daniele, MD, Medical Doctor, Santa Maria della Misericordia Rovigo Hospital
Organization: Santa Maria della Misericordia Rovigo Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2997CESC
Record Dates: First submitted 2021-10-11; First posted 2021-11-09 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Comparison of 3D Visualization and Microscope for VR Surgery
Keywords: Ngenuity; VR Surgery; Pucker; Macular Hole
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: Dual-arm, pilot, randomized, prospective, descriptive and comparative clinical study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control arm (Active Comparator): patients aﬀected by macular pucker or macular hole, whose internal limiting membrane peeling is performed using a traditional optical microscope (Leica F40)
  Interventions: Device: Macular surgery with standard operating microscope
- Experimental arm (Experimental): patients aﬀected by macular pucker or macular hole whose internal limiting membrane peeling is performed by 3D heads-up microscopy system (NGenuity 3D)
  Interventions: Device: Macular surgery with NGENUITY surgical display system

INTERVENTIONS:
Device: Macular surgery with NGENUITY surgical display system — Patient undergoes VR surgery with visualization using heads up display 3D monitor viewed by the operating surgeon
  Arms: Experimental arm
Device: Macular surgery with standard operating microscope — Patient undergoes VR surgery with visualization using standard operating microscope
  Arms: Control arm

SUMMARY:
Randomized, prospective, descriptive and comparative clinical study. The comparison is between a group of patients affected by macular pucker or macular hole, whose macular peeling is performed using a traditional optical microscope (Leica F40) - control arm, and a group of patients affected by macular pucker or macular hole whose macular peeling is performed by 3D heads-up microscopy system (NGenuity 3D, Alcon) - experimental arm.

It is a blind study for both the operator that collects data and for the statistician.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by macular pucker or macular hole, whose internal limiting membrane peeling need to be performed
* Willing and able to understand and sign an informed consent
* Willing and able to undergo postoperative examinations of the protocol program:
* ≥ 21 years of age, of both sexes and any race

Exclusion Criteria:

* History of ocular trauma or amblyopia.
* Other ocular pathologies (glaucoma, uveitis, diabetic retinopathy, diabetic macular edema, macular degeneration, Irvine Gass Syndrome, degenerative myopia, malformation of the optic disc, i.e.: tilted disc, optic disc pit, posterior staphyloma)
* Multiple procedures programmed during the surgery
* Pregnancy, lactation or programmed pregnancy during the course of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
SANFL detection | 2 weeks after surgery
  Post-surgical analysis of SANFL (Swelling of the Arcuate Nerve Fiber Layer) measured on infrared, blue auto-fluorescence images and OCT images of peripapillary region

SECONDARY OUTCOMES:
Intraoperative time | during surgery
  Mean duration of the surgical procedure
ILM staining | during surgery
  Number of internal limiting membrane staining procedures necessary
ILM grasping | during surgery
  Number of ILM grasping attempts.
Light | during surgery
  Lumen of light used
Surgeon ergonomics | during surgery
  Number of episodes of both back and neck pain
BCVA | baseline, 1 month and 3 months after surgery
  Best Corrected Visual Acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Maria della Misericordia Hospital, Rovigo, Italy

IPD SHARING:
Plan to Share IPD: Undecided